CLINICAL TRIAL: NCT00682916
Title: CCRC: FBCx® And Body Weight Regulation in Overweight Humans
Brief Title: Compare Effects of a Soluble Fiber on Weight and Blood Cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 200715061
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Obesity
Keywords: Obesity; Diabetes; Soluble Fiber; Overweight
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Subjects will fast prior to the initial visit. Subjects' weight, blood pressure and heart rate will be recorded, waist and hip circumferences measured, and body composition determined. They will receive either the soluble fiber or placebo tablets, in a coded bottle. They will be instructed to take 2 tablets per fat containing meal, 3 times a day within one hour of consuming the meal. They will also be asked to keep records of missed doses and any gastrointestinal symptoms (e.g.: heartburn, indigestion, diarrhea, constipation). During the 4th week, they will be asked to record food intakes for 3 days.
  After taking the supplement for 4 weeks, the participants will return to the clinic after an overnight fast. During this visit, they will turn in their 3-day dietary record. The studies performed during the initial baseline visit will be repeated. At this visit they receive the alternate supplement (placebo or active tablets) in a identical-looking coded bottle.
  Interventions: Dietary Supplement: Y288
- 2 (Placebo Comparator): Subjects will fast prior to the initial visit. Subjects' weight, blood pressure and heart rate will be recorded, waist and hip circumferences measured, and body composition determined. They will receive either the soluble fiber or placebo tablets, in a coded bottle. They will be instructed to take 2 tablets per fat containing meal, 3 times a day within one hour of consuming the meal. They will also be asked to keep records of missed doses and any gastrointestinal symptoms (e.g.: heartburn, indigestion, diarrhea, constipation). During the 4th week, they will be asked to record food intakes for 3 days.
  After taking the supplement for 4 weeks, the participants will return to the clinic after an overnight fast. During this visit, they will turn in their 3-day dietary record. The studies performed during the initial baseline visit will be repeated. At this visit they receive the alternate supplement (placebo or active tablets) in a identical-looking coded bottle.
  Interventions: Dietary Supplement: Y288

INTERVENTIONS:
Dietary Supplement: Y288 — Subjects will take 2 tablets per fat containing meal, 3 times a day, within one hour of consuming the meal
  Other Names: FBCx®
  Arms: 1
Dietary Supplement: Y288 — Subjects will take 2 tablets per fat containing meal, 3 times a day, within one hour of consuming the meal
  Other Names: FBCx®
  Arms: 2

SUMMARY:
Obesity and type 2 diabetes have clearly been linked together and identified as epidemics in much of the developed world. Historically several different dietary fibers have been used as means of reducing body weight and the related development of type 2 diabetes. These studies have generated mixed, if not inconsistent, results suggesting that none of these fibers promise a solution to either of these two conditions. We are proposing to investigate the effects of including a new soluble fiber, a-cyclodextrin, FBCx® (to be called Y288 in this study), into the diet of adult overweight volunteers.

DETAILED DESCRIPTION:
The overall aim is to investigate the effectiveness of a soluble dietary fiber, FBCx®, on weight loss and/or weight management, and blood lipid levels in overweight humans.

ELIGIBILITY:
Inclusion Criteria:

* 30 men and 30 women
* Age 18- 65 years
* BMI 25.0 - 32.0 Kg/m²
* fasting glucose <126 mg/dL
* Blood pressure < 140/85 mm Hg. Hypertension on stable drug regimen using 2 or fewer antihypertensives will be acceptable.
* Total plasma cholesterol <240 mg/dl, LDL-cholesterol <160 and triglycerides <400 mg/dl. Hyperlipidemia on a stable medication regimen using single anti-hyperlipidemic drug acceptable.

Exclusion Criteria:

* Pregnant women, women who plan to become pregnant during the study period
* Women who have given birth within the previous 12 months
* Lactating women
* History or presence of Type 2 diabetes; kidney disease; (creatinine >1.4); liver disease (X2 fold increase in AST or ALT); gout; cancer; untreated thyroid disease; gastrointestinal disease; other metabolic diseases or malabsorption syndromes
* Habitual low-fat intake (less than 20%)
* History of eating disorder
* Subjects who have lost 10% of body weight within the last 12 months or who plan to initiate a weight loss program
* Use of prescription or over-the counter anti-obesity medications or supplements (phenylpropanolamine, ephedrine, caffeine) for at least 6 months prior of study.
* Subjects with pacemakers will not participate in bioimpedance studies but will go through all the other testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
without any altering of dietary habits or exercise routine, individuals shall lose or maintain body weight during the active phase as compared to the placebo phase. | 4 weeks

SECONDARY OUTCOMES:
blood lipid levels during the active phase will be improved relative to the placebo phase. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sidika E Kasim-Karakas, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis, Sacramento, California, United States